CLINICAL TRIAL: NCT05652712
Title: A Real-World Study of Toripalimab in Chinese Patients With Lung Cancer(THUNDER Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Jiandong Zhang, Qianfoshan Hospital, Qianfoshan Hospital
Other Study IDs: YXLL-KY-2022(80)
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — toripalimab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Immunotherapy Regimen: Patients receiving different treatment regimens of Toripalimab in each center were consecutively enrolled from January 1, 2019 to December 31, 2022
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Toripalimab injection, recommended dose is 3 mg/kg, intravenous infusion every 2 weeks or 240 mg fixed dose, intravenous infusion every 3 weeks.
  Other treatment options are individualized according to the diagnosis and treatment experience of doctors in each center, diagnosis and treatment specifications and individual conditions of patients.

SUMMARY:
Our project is going to clarify the efficacy and safety of Toripalimab in lung cancer in the real world, and to evaluate the incidence of adverse events (AEs) of special interest during Toripalimab immunotherapy.

DETAILED DESCRIPTION:
Tumor immunotherapy, as another important treatment after surgical treatment, chemoradiotherapy and targeted therapy, has achieved great success and gradually become one of the standard treatment methods for tumors. Toripalimab is the first Chinese PD-1 inhibitor approved for the treatment of nasopharyngeal carcinoma, malignant melanoma, urothelial carcinoma, esophageal squamous cell carcinoma and non-small cell lung cancer. It has been widely used in clinical practice. Several clinical studies have confirmed that it is safe and effective. In recent years, several clinical studies have reported that Toripalimab alone or in combination can improve the response rate of cancer treatment and improve survival. The results of Toripalimab research are mainly derived from rigorously designed randomized controlled trials (RCTs), and the efficacy and safety in the real world still need to be further explored. Real world studies, based on a large sample size, non-randomly select treatment measures according to the actual condition and wishes of patients, and pay attention to meaningful outcome treatment, which is closer to real clinical practice, without extrapolation difficulties, and has more clinical practical value. Therefore, it is of great significance to carry out a real-world study to investigate the differences in the efficacy and adverse reactions of Toripalimab immunotherapy in Chinese lung cancer patients in order to better guide clinical practice, which also provides research direction and data support for further prospective studies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Cytologically or histologically confirmed lung cancer.
* Complete clinical data.
* Indications for immunotherapy with Toripalimab.

Exclusion Criteria:

* Lack of patient key data.
* Refusal or uncooperation with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive lung patients treated with Toripalimab
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival(OS) | 2 years
  OS was calculated from the date of randomization to death from any cause.

SECONDARY OUTCOMES:
Progression Free Survival(PFS) | 2 years
  PFS was defined as the time from the first day of study treatment to the first documented disease progression per irRC or death due to any cause, whichever occurred first.
Overall Response Rate (ORR) | 1 year
  ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR; disappearance of all target lesions) or Partial Response (PR; at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters).
Disease Control Rate(DCR) | 1 year
  The percentage of cases with remission (PR + CR) and stable lesions (SD) after treatment was assessable.
Health-related quality of life (HRQoL) | Within 1 year after starting Toripalimab treatment
  HRQoL measured by standardized EORTC questionaires (EORTC QLQ-C30)

OTHER OUTCOMES:
Number of Participants Experiencing Adverse Events (AEs) and serious adverse events (SAEs) | 1 year
  Adverse events are defined as any adverse medical events that occur in the participants taking the drugs and do not necessarily have a causal relationship with the treatment. AEs/SAEs were evaluated using NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China